CLINICAL TRIAL: NCT02871934
Title: Clinical Safety and Efficacy of Pharmacogenetics in Veteran Care
Brief Title: Integrating Pharmacogenetics In Clinical Care
Acronym: I-PICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SPLC-006-15S; IK2CX001262 (NIH)
Record Dates: First submitted 2016-08-16; First posted 2016-08-18 (Estimated); Results first posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Disease
Keywords: Pharmacogenetics; SLCO1B1 protein, human; OATP1B1 protein, human; Simvastatin; Cardiovascular disease; Cholesterol; Statin-related myotoxicity; Veterans; Point-of-care
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PGx+ (Experimental): Patients in the PGx+ (intervention) arm will have their SLCO1B1 results reported to their ordering provider immediately.
  Interventions: Genetic: SLCO1B1 Genotype
- PGx- (Experimental): Patient in the PGx- (control) arm will have their SLCO1B1 results reported to their ordering provider at the end of the study (after 12 months).
  Interventions: Genetic: SLCO1B1 Genotype

INTERVENTIONS:
Genetic: SLCO1B1 Genotype — Polymerase chain reaction (PCR) assay for SLCO1B1 rs4149056, with possible results T/T, T/C, or C/C.
  Other Names: SLCO1B1 Pharmacogenetic Test

SUMMARY:
This study will determine whether using a genetic test (for the SLCO1B1 gene) can help patients and providers choose the right type and dose of cholesterol-lowering statin medications to lower the risk of cardiovascular disease, while minimizing the muscle pain side effects that sometimes occur with statins.

DETAILED DESCRIPTION:
Variants at rs4149056 in the SLCO1B1 gene are associated with a greater risk of simvastatin-related myopathy. Despite the growing implementation of SLCO1B1 rs4149056 genotyping in health systems across the United States, there is little randomized controlled trial data on the impact of SLCO1B1 testing on clinical outcomes. The IPICC Study will use a randomized design to determine the impact of the clinical integration of SLCO1B1 genotype testing on important patient outcomes, including statin prescribing, LDL cholesterol, and statin-related myopathy. In addition, by enrolling statin-naive patients with a recent cholesterol panel, this trial will capture a moment of clinical decision-making when SLCO1B1 rs4149056 genotype might be most clinically relevant. This randomized-control trial has two primary aims:

Aim 1 (Drug safety): To determine the impact of SLCO1B1 pharmacogenetic testing on concordance with Clinical Pharmacogenetics Implementation Consortium (CPIC) pharmacogenetic guidelines for safe simvastatin prescribing and on the incidence of statin-related myopathy in VA (drug safety).

Aim 2 (Cardiovascular disease, CVD, prevention): To determine the impact of SLCO1B1 pharmacogenetic testing on LDL cholesterol levels and concordance with CVD prevention guidelines.

The I-PICC Study is enrolling 408 statin-naive primary care and women's health patients across the Veteran Affairs Boston Healthcare System. Eligible patients are aged 40-75 and have elevated risk of cardiovascular disease (CVD) according to American College of Cardiology/American Heart Association (ACC/AHA) guidelines. Primary care providers (PCPs) are also research subjects and consent via electronic health record (EHR) alerts. To model pharmacogenotyping at the point of care, the investigators are enrolling patients with recent cholesterol results when their PCPs order laboratory testing, indicating a moment of clinical decision-making about CVD risk. Enrolled patients are randomized to have their PCPs receive results through the EHR immediately (PGx+) vs. after 1 year (PGx-). The investigators will query clinical and pharmacy data for 1-year outcomes: myopathy and concordance with CPIC simvastatin guidelines (drug safety) and cholesterol levels and concordance with ACC/AHA guidelines (CVD risk reduction).

ELIGIBILITY:
Inclusion Criteria:

Providers:

* All providers in Primary Care and Women's Health at VA Boston Healthcare System will be eligible to participate.

Patients:

* Aged 40-75 years
* Have no history of statin use
* Have received VA care for at least the prior 6 months
* Are a patient of an enrolled provider
* Meet at least 1 of the following criteria:

  * cardiovascular disease (CVD)
  * diabetes
  * LDL cholesterol value >= 190 mg/dL
  * 10-year CVD risk of 7.5%, calculated with the ACC/AHA 2013 pooled risk equations

Exclusion Criteria:

* Patients will be ineligible if they:

  * Do not meet the inclusion criteria
  * Pregnant
  * Incarcerated or institutionalized

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Vassy, MD MPH, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vassy JL, Brunette CA, Majahalme N, Advani S, MacMullen L, Hau C, Zimolzak AJ, Miller SJ. The Integrating Pharmacogenetics in Clinical Care (I-PICC) Study: Protocol for a point-of-care randomized controlled trial of statin pharmacogenetics in primary care. Contemp Clin Trials. 2018 Dec;75:40-50. doi: 10.1016/j.cct.2018.10.010. Epub 2018 Oct 24. PMID 30367991
- [Result] Vassy JL, Gaziano JM, Green RC, Ferguson RE, Advani S, Miller SJ, Chun S, Hage AK, Seo SJ, Majahalme N, MacMullen L, Zimolzak AJ, Brunette CA. Effect of Pharmacogenetic Testing for Statin Myopathy Risk vs Usual Care on Blood Cholesterol: A Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2027092. doi: 10.1001/jamanetworkopen.2020.27092. PMID 33270123
- [Derived] Brunette CA, Miller SJ, Majahalme N, Hau C, MacMullen L, Advani S, Ludin SA, Zimolzak AJ, Vassy JL. Pragmatic Trials in Genomic Medicine: The Integrating Pharmacogenetics In Clinical Care (I-PICC) Study. Clin Transl Sci. 2020 Mar;13(2):381-390. doi: 10.1111/cts.12723. Epub 2019 Dec 18. PMID 31808996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PGx+ | PGx-
Started | 193 | 215
Completed | 193 | 215
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PGx+ | PGx- | Total
Number analyzed (Participants) | 193 | 215 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.8) | 63.9 (7.7) | 64.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 184 | 199 | 383
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 187 | 208 | 395
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 25 | 50
  White | 156 | 185 | 341
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 193 | 215 | 408
Smokers [Count of Participants; unit: Participants] | 59 | 78 | 137
Meeting ACC/AHA Criteria for Statin Therapy [Count of Participants; unit: Participants] — Categories sum to greater than 100% because criteria are not mutually exclusive. Abbreviations: ACC/AHA, American College of Cardiology / American Heart Association; ASCVD, atherosclerotic cardiovascular disease; LDL-C, low-density lipoprotein cholesterol.
  Participants
    ASCVD | 52 | 46 | 98
    LDL-C > 190 mg/dL | 5 | 6 | 11
    Diabetes | 47 | 51 | 98
    10-year ASCVD risk >= 7.5% | 171 | 196 | 367
SLCO1B1 Genotype [Count of Participants; unit: Participants]
  Normal function (T/T) | 148 | 140 | 288
  Decrease function (T/C) | 40 | 70 | 110
  Poor function (C/C) | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: 12-Month Change in LDL Cholesterol
Description: The primary CVD prevention outcome is 12-month change in low-density lipoprotein (LDL) cholesterol, defined as LDL value at 12 months minus LDL value at baseline.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | PGx+ | PGx-
Number analyzed (Participants) | 193 | 215
mg/dL | -1.1 (1.2) | -2.2 (1.3)

2. Secondary Outcome: Number of Participants With an American College of Cardiology/American Heart Association (ACC/AHA) Guideline Concordant Statin Prescription at 12 Months
Description: In 2013, the ACC/AHA endorsed guidelines that recommended prescribing statins of specific intensities (moderate or high) for distinct populations. Using patient characteristics and prescription data, the investigators will generate a 2-level CVD prevention outcome (concordant vs. non-concordant) for each participant, a measure of whether a patient's statin prescription is adequate for his/her level of CVD risk.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PGx+ | PGx-
Number analyzed (Participants) | 193 | 215
Participants | 12 | 14

3. Secondary Outcome: Number of Participants With Chart Review Documented Statin-related Myotoxicity at 12 Months
Description: Chart review of all patient notes during the 12 months after enrollment will be used to determine the proportion of patients in each arm who experienced statin-related muscle side effects during the observation period.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PGx+ | PGx-
Number analyzed (Participants) | 193 | 215
Participants | 2 | 3

4. Secondary Outcome: Number of Participants Meeting Clinical Pharmacogenetics Implementation Consortium (CPIC) Guidelines for Safe Simvastatin Prescription at 12 Months
Description: Clinical Pharmacogenetics Implementation Consortium (CPIC) guidelines recommend specific simvastatin doses when a patient's SLCO1B1 genotype is known. The investigators will compare each patient's medication prescriptions one year after enrollment to this guideline to generate a 2-level safety outcome (potentially safe vs. potentially unsafe simvastatin prescription) for each participant.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PGx+ | PGx-
Number analyzed (Participants) | 193 | 215
Participants | 193 | 215

5. Other Pre Specified Outcome: Participant Response Distributions to Belief in Medications Questionnaire at 12 Months
Description: Assessed by phone survey 12 months after enrollment. Consists of 2 items: "Do you agree or disagree with these statements?: "My health in the future will depend on my medicines" and "Medicines do more harm than good."
Time Frame: 12 months
Population: Data analyzed only for patients who completed the 12-month end-of-study survey.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx+ | PGx-
Number analyzed (Participants) | 169 | 203
Participants
  "My health in the future will depend on my medicines.": number analyzed (Participants) | 168 | 203
  "My health in the future will depend on my medicines.": Strongly agree | 28 | 30
  "My health in the future will depend on my medicines.": Agree | 65 | 84
  "My health in the future will depend on my medicines.": Uncertain | 29 | 37
  "My health in the future will depend on my medicines.": Disagree | 29 | 40
  "My health in the future will depend on my medicines.": Strongly disagree | 17 | 12
  "Medicines do more harm than good.": number analyzed (Participants) | 168 | 203
  "Medicines do more harm than good.": Strongly agree | 9 | 10
  "Medicines do more harm than good.": Agree | 26 | 20
  "Medicines do more harm than good.": Uncertain | 46 | 56
  "Medicines do more harm than good.": Disagree | 63 | 89
  "Medicines do more harm than good.": Strongly disagree | 24 | 28

6. Other Pre Specified Outcome: Number of Participants Recalling Pharmacogenetic Testing at 12 Months
Description: Assessed by phone survey 12 months after enrollment. Whether patient remembers receiving PGx results from provider and, if so, remembers the results and interpretation.
Time Frame: 12 months
Population: Result recall only assessed in intervention arm participants. Control participants received results 12 months after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx+
Number analyzed (Participants) | 169
Participants | 11

7. Other Pre Specified Outcome: Number of Participants Reporting Statin-related Muscle Side Effects at 12 Months
Description: Assessed by phone survey 12 months after enrollment. Whether patient attributes muscle pains, weakness, or cramps to a statin taken in the prior 12 months.
Time Frame: 12 months
Population: Data analyzed only for patients who completed the 12-month end-of-study survey.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx+ | PGx-
Number analyzed (Participants) | 169 | 203
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 12 months
Description: Mortality and adverse event data collected non-systematically due to minimal risk nature of the trial intervention. Most mortality events discovered when attempting to reach patient for end-of-study survey. Any participant death or adverse event discovered by study staff during the observation period or via attempts to make contact for end-of-study survey (per protocol, contacts occurred up to 3 months after end of 12-month observation period) data collection are reported.
Arm/Group | PGx+ | PGx-
All-Cause Mortality (participants affected / at risk) | 8/193 | 5/215
Serious Adverse Events (participants affected / at risk) | 0/193 | 0/215
Other Adverse Events (participants affected / at risk) | 0/193 | 0/215

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT02871934/Prot_SAP_000.pdf